CLINICAL TRIAL: NCT00432692
Title: Falls Prevention for People With Increased Risk of Fractures as a Result of Osteoporosis: a Randomized Controlled Study on the Effects of a Modified Program
Brief Title: Falls Prevention in Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMK001
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2007-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis; falls; prevention; elderly; exercise; incidence; obstacle avoidance
MeSH Terms: conditions — Osteoporosis; Motor Activity

INTERVENTIONS:
Procedure: Falls Prevention Program

SUMMARY:
The purpose of this study is to determine wether a falls prevention program can reduce fall incidence in people with osteoporosis.

DETAILED DESCRIPTION:
Falling is a major health problem in the elderly causing physical and psychosocial problems. People with osteoporosis are at higher risk for fractures due to falling, because of decreased bone strength. The 'Nijmegen Falls Prevention Program" (NFPP) (Weerdesteyn et al, 2006) has been shown to reduce fall incidence rates by 46% in healthy community-dwelling elderly. This program was adapted in order to meet the specific demands and constraints of people with osteoporosis.

The contents of the program are an obstacle course, walking exercises, the practice of fall techniques, adjustment of gait abnormalities, weight bearing exercises and educational sessions.

The effectiveness of the program will be evaluated in a randomized clinical trial. Primary outcome measure is fall incidence. Additionally, laboratory assessments of gait and obstacle avoidance will be conducted in conjunction with questionnaires about balance confidence and activity level.

ELIGIBILITY:
Inclusion Criteria:

* osteoporosis (DXA T-score < -2.5 in hip and/or vertebrae)
* able to walk at least 15 minutes without an helping device
* 65 years or older
* community dwelling
* at least one fall in the prior year

Exclusion Criteria:

* severe cardiac, pulmonary or musculoskeletal disorders
* pathologies associated with increased fall risks (i.e. stroke or Parkinson's disease)
* use of psychotropic drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fall incidence, which is measured by monthly fall registration cards

SECONDARY OUTCOMES:
Obstacle avoidance performance
Fear of falling (ABC)
Activity level (LAPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Smulders, MSc, Principal Investigator — Sint Maartenskliniek; Vivian Weerdesteyn, PhD, Principal Investigator — Sint Maartenskliniek; Wim van Lankveld, PhD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Nijmegen, Netherlands

REFERENCES:
- [Derived] Smulders E, Weerdesteyn V, Groen BE, Duysens J, Eijsbouts A, Laan R, van Lankveld W. Efficacy of a short multidisciplinary falls prevention program for elderly persons with osteoporosis and a fall history: a randomized controlled trial. Arch Phys Med Rehabil. 2010 Nov;91(11):1705-11. doi: 10.1016/j.apmr.2010.08.004. PMID 21044715